CLINICAL TRIAL: NCT03447951
Title: A Phase II Study to Assess the Safety and Efficacy of PTS100 in Primary Hepatocellular Carcinoma Patients Who Are Ineligible for Operation or Current Locoregional Therapy
Brief Title: A Study of PTS100 in Primary HCC Patients
Acronym: OASES
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gongwin Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GW-020202
Record Dates: First submitted 2018-02-13; First posted 2018-02-27 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — 4-toluenesulfonamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PTS100 (Para-Toluenesulfonamide): 30%TTV (Experimental): Total dose = 30% total tumor volume
  Interventions: Drug: Para-Toluenesulfonamide

INTERVENTIONS:
Drug: Para-Toluenesulfonamide — A total dose of PTS100 in this study, the expected accumulated dose in the treatment duration, depends on the patient's tumour size. For each patient, up to 4 tumors, each not exceeding 8.8 cm in diameter, are selected for treatment by the joint decision of the investigator and the radiologist. The total dose is defined as the accumulated dose in treatment duration. The total dose is assigned as 30% of TTV for each patient and maximum TTV should be less than 366 cm3.
  Other Names: PTS100

SUMMARY:
This study is being performed to evaluate the efficacy and safety of 30% PTS100 of total tumor volume as intra-tumoral injection therapy in primary Hepatocellular Carcinoma patients who are ineligible for operation or local regional therapy.

DETAILED DESCRIPTION:
BCLC stage B patients who are ineligible for operational or current locoregional therapy. Enrolled patients are assigned to 30% of total tumor volume. PTS100 is administrated via intratumoral injection. The required total dose is given in separate injection days, with maximal daily dose up to 10 mL at first IP administration, and is adjusted based on each patient's tolerability along the treatment. The treatment course lasts up to completion of the total dose, and the efficacy is evaluated 28 days afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥ 20 years and ≤ 80 years of age.
* Patients with clinically confirmed primary HCC following American Association for the Study of Liver Diseases (AASLD, Appendix 1) guidance:

  1. Cyto-histological evidence, or
  2. Coincident imaging evidence using computerized tomography (CT) or magnetic resonance imaging (MRI)
* Based on investigator discretion, patients who are diagnosed at Barcelona Clinic Liver Cancer (BCLC) stage B and are ineffective or unsuitable for resection, immediate liver transplantation, Trans Arterial Chemoembolization (TACE), or current local ablative treatment and meet all of the following conditions at study entry:

  1. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
  2. Child Pugh score class A or B.
* Patients with at least one measurable lesion with size ≥ 1 cm.
* Patients with cumulative total treated tumor volume ≤ 366 cm3 and ≤ 4 target tumors.
* Patients with adequate bone marrow, liver and renal function within 28 days prior to study entry, as defined by the following:

  1. Hemoglobin > 10.0 g/dl.
  2. Absolute neutrophil count (ANC) > 1,500/mm3.
  3. Platelet count > 80k/mm3 correctable by component therapy.
  4. Albumin ≥ 3 g/dl.
  5. Total bilirubin < 2 mg/dL.
  6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 5 x upper normal limit (UNL).
  7. Blood urea nitrogen (BUN) and serum creatinine < 1.5 x UNL.
  8. International normalized ratio (INR) < 1.5 or prothrombin time (PT) < 15 seconds.
* Patients with life expectancy > 3 months as judged by investigator.
* Patients who understand and comply to the study procedure and be willing to provide a written informed consent form.

Exclusion Criteria:

* Infiltrative HCC or tumor burden ≥ 50% of liver parenchyma.
* Patients with cumulative total treated tumor volume > 366 cm3 or more than 4 target tumors.
* Any target tumor exceeds 8.8 cm in diameter.
* The treated tumor is located in close proximity to another organ (e.g. gall bladder, liver capsule, diaphragm ) or major blood vessel and less than 0.5 cm in distance .
* Presence of metastasis or vascular invasion.
* Systemic chemotherapy treatment for HCC within 12 weeks prior to study entry.
* Major surgery within 4 weeks prior to study entry (e.g. thoracolaparotomy is not allowed, but noninvasive surgery, e.g. biopsy, is allowed).
* Use of any investigational drugs, biologics, or devices within 4 weeks prior to study entry or planned use during the course of study.
* Any other severe disease (e.g. active infection, uncontrolled diabetes mellitus, severe heart dysfunction or angina, gastric ulcer, active auto-immune disease) judged by the investigator to limit subject participation in the study.
* Female subjects who are pregnant or lactating. Women of childbearing potential must have a negative urine pregnancy test performed within seven days prior to the start of study drug and agree to practice medically acceptable contraceptive regimen from screening until at least 28 days after the study treatment. Patients who are postmenopausal for at least 1 year (> 12 months since the last menstrual cycle) or were surgically sterilized do not require the pregnancy test.
* Known or suspected allergy and/or hypersensitivity to any of the ingredients of PTS100.
* Any target lesion blocked by bile ducts or important blood vessels, judged by investigator, that is difficult to conduct intratumoral injection.
* Any condition, judged by investigator, that shows subjects are not suitable for participation.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2018-06-19 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 4-week post treatment
  To evaluate the efficacy, measured by objective response rate (ORR) of pooled treatment groups based on the modified RECIST (mRECIST) criteria at concluding visit.

SECONDARY OUTCOMES:
Local disease control rate (LDCR) | 4-week post treatment
  Local disease control rate (LDCR) of pooled treatment groups based on the modified RECIST (mRECIST) criteria at concluding visit.
Time to treated tumor progression (TTTTP) | 4-week post treatment, then every 2 months follow up with imaging will be continued for 12 months
  Time to treated tumor progression (TTTTP) of pooled treatment groups
Three-year overall survival (OS) | Time from first IP administration to patient death or to the date of 3 years after first IP administration
  Three-year overall survival of pooled treatment groups
Time to tumor stage progression (TSP) | Time from first IP administration to every 2 months follow up with imaging will be continued for 12 months
  Time to tumor stage progression of pooled treatment groups
Difference in ORR between group 1 and group 2 | 4-week post treatment
  Difference in ORR between 20% group and 30% group at concluding visit
Difference in LDCR between group 1 and group 2 | 4-week post treatment
  Difference in LDCR between 20% group and 30% group at concluding visit
Difference in TTTTP between group 1 and group 2 | 4-week post treatment to every 2 months follow up with imaging will be continued for 12 months
  Difference in TTTTP between 20% group and 30% group at concluding visit
Incidence of Treatment-Emergent Adverse Events | Enrollment to 4-week post treatment
  Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v4.0
FACT-Hep quality of life score | 4-week post treatment and every 2 months follow up will be continued for 12 months
  To evaluate the health-related Quality of life, assessed by change in Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep, version 4, Traditional Chinese). The FACT-Hep, version 4, Traditional Chinese Scale is a patient completed questionnaire consisting 45 items that assesses health related quality of life (HRQL) in HCC patients. The FACT-Hep, version 4, Traditional Chinese consists of the 27-item FACT-G assessing generic HRQL concerns and 18-item Hepatobiliary Subscale assessing disease-specific issues. Instrument scoring yields a range from 0 to 180 with higher scores representing better patient status. This questionnaire should be completed by patient prior to any procedures being performed at the visit, if possible. The form should then be checked by site staff for completeness.
EQ-5D-5L quality of life score | 4-week post treatment and every 2 months follow up will be continued for 12 months
  To evaluate the health-related Quality of life, assessed by change in EuroQol 5 dimensions 5 level (EQ-5D-5L). It comprises the same 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels. However, this results have no arithmetic properties and should not be used as a cardinal score. This questionnaire should be completed by the patient prior to any procedure being performed at the visit, if possible. The form should then be checked by site staff for completeness.

CONTACTS AND LOCATIONS:
Overall Officials: Ja Der Liang, Principal Investigator — National Taiwan University Hospital
Locations (3):
- Taiwan (3):
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei